CLINICAL TRIAL: NCT05671471
Title: Accidental Reactions in a French Cohort of Children With Peanut and/or Tree Nut Allergy.
Brief Title: Accidental Reactions in Peanut/Tree Nut Allergic Children
Acronym: ALLERGY
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0099; 2021-A00746-35 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2022-11-03; First posted 2023-01-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Peanut and Tree Nut Allergy
Keywords: Peanut allergy; tree nut allergy; peanut immunotherapy; anaphylaxis; real life
MeSH Terms: conditions — Nut and Peanut Hypersensitivity; Peanut Hypersensitivity; Nut Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allergic Children: Patients followed in the Pediatric Allergy and Pulmonology Unit, CHU Lille, aged 0-18 years with peanut and/or tree nut allergy

SUMMARY:
Food allergy is an immune reaction, triggered by food protein allergens, of varying severity, from mild local reaction to life threatening anaphylaxis and fatalities.

Peanut is a plant from the botanical family of the Fabaceae, more commonly known as legumes. The prevalence of peanut and tree nut allergy is increasing. In France (ELFE cohort), it is estimated to 0.93%. The tree nuts include mainly almond, hazelnut, pistachio, cashew nut, walnut, pecan nut and Brazil nut. Allergy's prevalence is estimated to 0.54% in children up to 5.5 years. Peanut allergy is a main cause of anaphylaxis and deaths due to food allergy.

Recurrence of food allergy is a main concern. The risk has been estimated to 10% per year for peanut.

In France, Data in real-life on the rate of recurrence of allergic reactions and anaphylaxis to peanut/tree-nut as well as risk factors, are lacking.

The objective of this study is to assess the frequency of allergic reaction to peanut and tree-nuts, to describe the reactions' characteristics and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed allergy to peanuts and/or nuts

Exclusion Criteria:

* Other chronic diseases, except allergic comorbidities (asthma, rhinitis, atopic dermatitis, other food allergy)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients followed in the Pediatric Allergy and Pulmonology Unit, CHU Lille, aged 0-18 years with peanut and/or tree nut allergy
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
the number of episode of allergic reactions in real life | At 1 year

SECONDARY OUTCOMES:
the severity of the allergic reactions according to a validated scale (FASS scale) | At 1 year
interview for the characteristics of the allergic reactions | At 1 year
  the characteristics of the reactions: symptoms, triggering food and quantity, location, emergency kit available, treatment administered, evolution (hospitalization or emergency room)
interview to defined the risks factor associated | At 1 year
  risk factors for reaction:
  * Other known allergies
  * Asthma
  * Atopic dermatitis
  * Allergic rhinoconjunctivitis
  * Patient characteristics: sex, age

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DESCHILDRE, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France